CLINICAL TRIAL: NCT03671850
Title: A Phase 2 Study to Evaluate the Efficacy and Safety of Postremission Therapy Using VT-EBV-N in EBV Positive Extranodal NK/T Cell Lymphoma Patients
Brief Title: VT-EBV-N for Treatment of Severe in EBV Positive Extranodal NK/T Cell Lymphoma Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ViGenCell Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VT-EBV-201
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-03

CONDITIONS: Extranodal NK/T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VT-EBV-N (Experimental): Epstein-barr virus human cytotoxic T lymphocytes (EBV-CTL)
  Interventions: Biological: VT-EBV-N
- Placebo (Placebo Comparator): Peripheral blood mononuclear cell, PBMC
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: VT-EBV-N — Epstein-barr virus human cytotoxic T lymphocytes (EBV-CTL)
  Arms: VT-EBV-N
Other: Placebo — Peripheral blood mononuclear cell, PBMC
  Arms: Placebo

SUMMARY:
The study aims to evaluate the efficacy and safety of VT-EBV-N (EBV-CTL) administration in ENKL patients after complete remission (CR). This is to prove the effect of VT-EBV-N (EBV-CTL) in prevention of ENKL relapse compared to placebo, by checking the primary endpoint of DFS rate (disease free survival, no relapse or death after randomization) at 2 years (103 weeks) for the last subject enrolled. 50% of the subjects will be administered VT-EBV-N (EBV-CTL), while the remaining subjects will be administered a placebo.

DETAILED DESCRIPTION:
NK/T-cell lymphoma is a malignant tumor originating in NK cells and T lymphocytes. ENKL is associated with Epstein-Barr virus (EBV) infection and typically occurs in the nasal area, being termed ENKL, nasal type.EBV is a common virus in the herpes family. EBV infection in patients with lowered immunity such as those with Acquired Immune Deficiency Syndrome or those taking immunosuppressants after bone marrow transplant may induce lymphoproliferative diseases or cancer.

VT-EBV-N (EBV-CTL) is a cytotoxicity T lymphocyte (CTL) targeting EBV expressed tumor cells indicated for ENKL. Antigen-presenting cells derived from the patient's own blood is used to activate T-cells in a test tube to recognize EBV, which are then expanded in vitro and infused into the patient's body. Targeted immunotherapy using EBV-CTL is a safe form of treatment that can improve long-term disease-free survival rates by boosting antitumor immunity without affecting other tissues apart from tumor cells.

ELIGIBILITY:
Inclusion Criteria:

1. EBV positive extranodal NK/T cell lymphoma (ENKL) patients pathologically confirmed according to WHO classification at first diagnosis
2. Patients whose complete remission (CR) has been confirmed within 6 months before screening and maintained, presenting high risk of relapse due to one or more of the following 1) Patients who are EBV detectable at initial diagnosis, with one or more of the following high risk factors 60 years of age or older, Ann Arbor stage II ~ IV, non-nasal type disease, local invasiveness (defined with T3 or T4), elevated LDH (> upper limit of normal)) 2) Patients confirmed to have EBV DNAemia (> 2000 copies/ml) during or after treatment 3) Patients who achieved remission from secondary or greater remission induction therapy after the failure of primary remission induction, or achieved remission after relapse
3. 19 years and above to 75 years and below
4. Patients with ECOG performance criteria score of 0 to 2
5. Patients with acceptable hematopoietic function (ANC ≥ 1.5 x 109 /L, PLT ≥ 100 x 109 /L, Hb ≥ 9 g/dL)
6. Patients with acceptable liver function (total bilirubin < 2 x upper limit of normal, AST/ALT < 3 x upper limit of normal)
7. Patients with renal function of eGFR > 50 or better
8. Patients with life expectancy of 6 or longer
9. Patients who have agreed to use two different types of birth control during the study period (Females of childbearing age or within 2 years after menopause have to show negative results in urine pregnancy test) (E.g., dual contraception using oral contraceptives, contraceptive implant, contraceptive injection, or contraceptive patch combined with intrauterine device, spermicide foam or gel, contraceptive film, vaginal diaphragm, cervical cap, condom, etc.)
10. Patients who have voluntarily given written consent to participate in this study

Exclusion Criteria:

1. Other pathological classifications of nasal cavity lymphoma than ENKL at initial diagnosis
2. Patients with ENKL that has invaded the central nervous system
3. Patients in PR, SD or PD state, not complete remission (CR)
4. Patients who cannot generate EBV-CTL
5. Patients who have received allogeneic stem cell transplantations
6. Patients with severe or uncontrolled medical disorders(diabetes exceeding HbA1C9%, severe hypertension exceeding 180/110 mmHg, heart failure of NYHA class Ⅲ or Ⅳ, myocardial infarction diagnosed within 6 months prior to screening)
7. Patients with apparent infection (HIV infection, chronic hepatitis B, chronic hepatitis C, active tuberculosis, etc.)
8. Patients with malignant tumors or previous history of malignant tumors except completely recovered non-melanoma skin cancer or stage 0 (in situ) cervical carcinoma
9. Patients currently receiving treatment for ENKL such as chemotherapy, hormone therapy, or immunotherapy
10. Patients with hypersensitivity to the investigational product or pretreatment products, including cryoprotectants

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-04-09 (Actual); Primary Completion 2023-12-04 (Estimated); Study Completion 2024-06-03 (Estimated)

PRIMARY OUTCOMES:
No relapse or death due to any reason after randomization | Randomization (8 weeks before administration) ~ 116 weeks after treatment period

SECONDARY OUTCOMES:
No death after randomization | Randomization (8 weeks before administration) ~ 116 weeks after treatment period
No relapse or death due to any reason after randomization | Randomization (116 weeks after treatment period) ~

CONTACTS AND LOCATIONS:
Overall Officials: Seok-Goo Cho, Principal Investigator — The Catholic University of Korea
Locations (8):
- South Korea (8):
  - Inje University Busan Paik Hospital, Busan
  - Keimyung University Daegu Dongsan Hospital, Daegu
  - Hallym Univ. Medical Center, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Seoul St.Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No